CLINICAL TRIAL: NCT04724005
Title: Project Affinity: Excess Cancer Blood Testing Technique
Brief Title: Project Affinity: Excess Cancer Blood Testing
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 289800
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No drug — No drug used

SUMMARY:
Study investigating cancer blood samples on an iterative measurement systme

ELIGIBILITY:
Inclusion Criteria:

* Undergoing SACT
* Routine blood tests

Exclusion Criteria:

* Not had first cycle of SACT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Above 18 years of age. Undergoing SACT treatment. Going to hospital for routine blood tests.
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Viability of measurement technique | 12 months
  Viability of measurement technique

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be decided